CLINICAL TRIAL: NCT06947304
Title: A Phase 1, Open-Label Study Evaluating the Effect of Miricorilant on Hepatic Lipids in Patients With Presumed Metabolic Dysfunction-Associated Steatohepatitis (MASH)
Brief Title: Evaluation of Miricorilant on Liver Fat in Patients With MASLD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Collaborators: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORT118335-858
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Nonalcoholic Steatohepatitis (NASH); Metabolic Dysfunction-Associated Steatohepatitis (MASH); Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD); Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: Nonalcoholic Fatty Liver Disease (NAFLD); Nonalcoholic Steatohepatitis (NASH); Metabolic dysfunction-Associated Steatohepatitis (MASH); Metabolic dysfunction-Associated Steatosis Liver Disease (MASLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Miricorilant- 100 mg (Experimental): Patients who meet the entry criteria for study CORT118335-858 will be enrolled to receive 100 mg of miricorilant every day for 6 weeks.
  Interventions: Drug: Miricorilant

INTERVENTIONS:
Drug: Miricorilant — 100 mg administered orally, once daily

SUMMARY:
A Phase 1, Open-Label Study Evaluating the Effect of Miricorilant on Hepatic Lipids in Patients with Presumed Metabolic Dysfunction-Associated Steatohepatitis (MASH)

DETAILED DESCRIPTION:
Approximately 8 patients who are eligible for participation in the study will be assigned to a single dose cohort receiving 100 mg of miricorilant daily. The total duration of participation for each patient is expected to be up to 16 weeks, comprising a 6-week screening period, a 6-week treatment phase, and a 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* AST > 17 U/L for women and AST > 20 U/L for men. The AST inclusion criterion does not apply to participants with an eligible historical liver biopsy performed within 12 months of screening showing one of the following:

  1. NAFLD Activity Score (NAS) ≥ 4 (with at least 1 point in each subcomponent of steatosis, inflammation, and ballooning) and NASH Clinical Research Network (CRN) fibrosis score of F0 OR
  2. NAS ≥ 3 (with at least 1 point in each subcomponent of steatosis, inflammation, and ballooning) and NASH CRN fibrosis score of F1 OR
  3. NAS ≥ 2 (with at least 1 point in subcomponent of ballooning or inflammation) and a NASH CRN fibrosis score of F2-3
* MRI-PDFF with ≥ 8% steatosis; this assessment must be performed within 4 weeks of the Baseline Visit.
* Presence of at least 1 of the following metabolic syndrome characteristics that increase the risk of MASH:

  a. Diagnosis of type 2 diabetes managed with diet alone or diet and metformin (metformin dose must be stable for at least 1 month prior to screening) OR b. Presence of 3 or more components of metabolic syndrome: i. Fasting blood glucose ≥ 100 mg/dL (5.6 mmol/L) or treatment for elevated blood glucose with metformin ii. Systolic blood pressure ≥ 130 mm Hg, diastolic blood pressure ≥ 85 mm Hg, or treatment for hypertension iii. Serum TG ≥ 150 mg/dL (1.7 mmol/L) iv. Serum high-density lipoprotein cholesterol (HDL) < 40 mg/dL (1 mmol/L) in men and < 50 mg/dL (1.3 mmol/L) in women or drug treatment for low HDL v. Having overweight or obesity (body mass index [BMI] ≥ 25 kg/m2 [BMI
  * 23 kg/m2 in Asians]), or increased waist circumference ≥ 102 cm (40 in) in men and ≥ 88 cm (35 in) in women (men ≥ 90 cm [35.4 in]; women ≥ 80 cm [31.5 in] in Asians).

Other inclusion criteria may apply

Exclusion Criteria:

* Participation in another clinical trial for MASH or weight loss (e.g., GLP-1 receptor agonists) within the last 3 months.
* Participation in any other clinical trial within the last 3 months or 5 half-lives of the treatment, whichever is longer.
* Women who are pregnant, planning to become pregnant, or lactating.
* BMI < 18 kg/m² or > 45 kg/m².
* Significant alcohol consumption exceeding 20 g/day for women or 30 g/day for men within 1 year prior to screening.
* Positive urine drug screen for amphetamines, cocaine, opiates, or cannabinoids.
* Known or suspected cirrhosis or signs of hepatic decompensation.
* Other chronic liver diseases such as hepatitis B or C, autoimmune hepatitis, primary biliary cholangitis, or Wilson's disease.
* History of myocardial infarction, unstable angina, or stroke within 3 months prior to screening.
* Uncontrolled hypertension (systolic > 160 mm Hg or diastolic > 100 mm Hg).
* Current use of medications prohibited due to potential drug-drug interactions with study treatment.
* Contraindications to magnetic resonance imaging (MRI).

Other exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in fasting hepatic lipogenesis after 6 weeks of treatment | Baseline to Week 6
Change in peak lipogenesis after 6 weeks of treatment. | Baseline to Week 6

SECONDARY OUTCOMES:
Change in liver fat content by MRI-PDFF after 6 weeks of treatment | Baseline to week 6

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Juneja, MD, Study Director — Corcept Therapeutics
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No